CLINICAL TRIAL: NCT01537289
Title: A Prospective Randomized Study of 14-French (14F) Pigtail Catheters Versus 28F Chest Tubes in Patients With Traumatic Pneumothorax: Impact on Tube-Site Pain and Failure Rate
Brief Title: Pigtail Catheter Versus Chest Tube in the Management of Traumatic Pneumothorax
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Arizona (Other)
Responsible Party: Principal Investigator, Narong Kulvatunyou, Assistant Professor, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10-0405-03
Record Dates: First submitted 2012-02-09; First posted 2012-02-23 (Estimated); Last update posted 2012-02-23 (Estimated); Status verified 2012-02

CONDITIONS: Traumatic Pneumothorax
Keywords: Trauma; Pneumothorax
MeSH Terms: conditions — Wounds and Injuries; Pneumothorax | interventions — Chest Tubes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pigtail catheter (Experimental)
  Interventions: Device: Pigtail catheter insertion (Cook)
- Traditional chest tube (Active Comparator): 28-French chest tube
  Interventions: Device: chest tube (28-French)

INTERVENTIONS:
Device: Pigtail catheter insertion (Cook) — insertion of pigtail catheter to decompress pneumothorax
  Other Names: Cook Critical Care, Cook Incorporated, Bloomington, IN)
  Arms: Pigtail catheter
Device: chest tube (28-French) — inserting chest tube to decompress pneumothorax
  Other Names: 28-French chest tube
  Arms: Traditional chest tube

SUMMARY:
A small 14-French(F) pigtail catheter (PC) has been shown to work equally well with traditional 32-40F chest tube (CT), especially in traumatic pneumothorax.

There are no clinical data on tube-site pain. The investigators hypothesize that PC tube site pain is less than CT.

DETAILED DESCRIPTION:
Primary outcome: - Tube site pain

* Pain medication requirement

Secondary outcome: failure rate insertion-related complication

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and above
* Suffer traumatic pneumothorax that requires chest tube insertion

Exclusion Criteria:

* Emergency chest tube insertion
* patient refuses
* patient is unable to provide or rate pain assessment
* prisoner
* pregnancy
* patient with GCS less than 13

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2010-07; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
Change in Tube-site pain, pain medication requirement | day 0, 1, 2

SECONDARY OUTCOMES:
failure rate | patients will be followed for the duration of hospital stay, an expected average of 2 weeks
Insertion-related complication | day 0

CONTACTS AND LOCATIONS:
Overall Officials: narong kulvatunyou, MD, Principal Investigator — University of Arizona
Locations (1):
- University of Ariznoa Medican Center, Main campus, Tucson, Arizona, United States

REFERENCES:
- [Derived] Kulvatunyou N, Erickson L, Vijayasekaran A, Gries L, Joseph B, Friese RF, O'Keeffe T, Tang AL, Wynne JL, Rhee P. Randomized clinical trial of pigtail catheter versus chest tube in injured patients with uncomplicated traumatic pneumothorax. Br J Surg. 2014 Jan;101(2):17-22. doi: 10.1002/bjs.9377. PMID 24375295